CLINICAL TRIAL: NCT06769672
Title: The Effect of Dual-task Training Combined With tDCS on Cognitive-motor Interference and Related Brain Activity in Stroke Patients
Brief Title: Dual-task Training Combined With tDCS on Cognitive-motor Performance and Brain Activity in Stroke Patients
Acronym: dual-task tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Marco PANG_tDCS
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Cortical Excitability
Keywords: Dual-task training; Cognitive-motor interference; tDCS
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS combined with dual-task group (Experimental): patients receive three active tDCS and three dual motor-cognitive exercise training per week for four weeks.
  Interventions: Other: active tDCS with dual-task training
- sham tDCS combined with dual-task group (Active Comparator): Patients receive three sham tDCS and three dual cognitive-motor exercise training per week for four weeks.
  Interventions: Other: sham tDCS with dual-task training

INTERVENTIONS:
Other: active tDCS with dual-task training — participants receive three 20-minute active tDCS treatment and three 60-minute COGMOTION dual-task exercise sessions per week for four consecutive weeks.
  Arms: active tDCS combined with dual-task group
Other: sham tDCS with dual-task training — participants receive three 20-minute sham tDCS treatment and three 60-minute COGMOTION dual-task exercise sessions per week for four consecutive weeks.
  Arms: sham tDCS combined with dual-task group

SUMMARY:
The purpose of this study is to evaluate tDCS combined with cognitive-motor training on dual-task interference during dual-task walking, dual-task foot pedaling and the corresponding alterations of brain activity.

DETAILED DESCRIPTION:
In China, the prevalence of stroke increased by 106.0% (93.7-118.8) between 1990 and 2019, highlighting the persistent and substantial burden of this condition. Post-stroke recovery, particularly the ability to achieve community ambulation, plays a critical role in improving health-related quality of life. Effective community ambulation in daily life requires the ability to dual-task-namely, to perform concurrent tasks requiring attentional resources while maintaining walking function and balance. Emerging evidence suggests that stroke survivors face greater challenges in walking function and dual-task balance compared to their age-matched, able-bodied counterparts. For instance, when tasked with recalling a shopping list while walking, stroke patients exhibit a more pronounced decline in both walking speed and cognitive performance relative to control groups. Given the necessity for stroke survivors to reintegrate into the community, it is imperative to thoroughly investigate this phenomenon of cognitive-motor interference.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of stroke, stroke onset of more than 6 months,
* aged 50 or more,
* capable of following verbal and visual instructions,
* having a Montreal Cognitive Assessment score ≥ 22,
* able to walk for 10 meters with/without a mobility aid,
* community-dwelling, unilateral stroke

Exclusion Criteria:

* neurological disorders, gait-precluding pain or comorbidity,
* receiving any formal rehabilitation training,
* contraindications to exercise (e.g., unstable angina),
* contraindications to fNIRS, MRI, and tDCS (e.g., brain skin injury, pacemaker, metal implants in the brain),
* history of seizure or epilepsy,
* color blindness.
* unable to walk with/without a mobility aid while responsing stimulus by the remote control

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dual-task gait speed | Through study completion, an average of 1 year
  Gait speed under dual-task condition will be recorded
Dual-task cognitive performance | Through study completion, an average of 1 year
  Number of correct responses will be measured during dual-task conditions

SECONDARY OUTCOMES:
Oxyhemoglobin concentration changes of the brain | Through study completion, an average of 1 year
  Oxyhemoglobin concentration changes will be measured using functional near infra-red spectroscopy during dual-task walking
Dual-task gait performance 1 | Through study completion, an average of 1 year
  Gait cadence will be measured during dual-task walking
Dual-task gait performance 2 | Through study completion, an average of 1 year
  Gait cycle duration will be measured during dual-task walking
Dual-task gait performance 3 | Through study completion, an average of 1 year
  Stride length will be measured during dual-task walking
Dual-task cognitive performance 1 | Through study completion, an average of 1 year
  Correct reaction time under dual-task walking will be recorded
Blood oxygenation level changes of the brain | Through study completion, an average of 1 year
  Blood oxygenation level changes will be measured using Magnetic Resonance Imaging during dual-task foot pedaling
Dual-task stride time | Through study completion, an average of 1 year
  cadence under dual-task foot pedaling will be recorded
Dual-task cognitive performance 2 | Through study completion, an average of 1 year
  Number of correct responses under dual-task foot pedaling will be recorded
Dual-task gait performance 4 | Through study completion, an average of 1 year
  Step time under dual-task walking will be recorded

OTHER OUTCOMES:
Dual-task peak angular velocity | Through study completion, an average of 1 year
  Peak angular (dorsi-plantar flexion) velocity under dual-task foot pedaling will be recorded
Dual-task cognitive performance 3 | Through study completion, an average of 1 year
  Correct reaction time under dual-task foot pedaling will be recorded
Single-task walking speed | Through study completion, an average of 1 year
  10-meter walking test will be used to assess single-task walking speed in meters per second
Balance 1 | Through study completion, an average of 1 year
  Mini Balance Evaluation Systems Test will be used to assess postural control, with total points from 0-28. Higher points indicate better performance.
Balance 2 | Through study completion, an average of 1 year
  Activities-specific Balance Confidence Scale will be used to assess confidence of functional balance performance, with total points from 0-100. Higher points indicate better performance.
Cognitive performance | Through study completion, an average of 1 year
  Stroop color word test will be used to assess executive function
Cognitive performance 1 | before the initiation of training
  Montreal Cognitive Assessment will be used to assess global cognition, with total points from 0-30. Higher points indicate better performance.
Cognitive performance 2 | Through study completion, an average of 1 year
  Trail Making Test will be used to assess executive function
Fall incidence | Through study completion, an average of 1 year
  Monthly telephone interviews for recording fall incidence
dual-task walking performance at maximal speed | Through study completion, an average of 1 year
  Walking time under dual-task walking at maximal speed will be recorded
dual-task cognitive performance at maximal speed | Through study completion, an average of 1 year
  Accuracy under dual-task walking at maximal speed will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR